CLINICAL TRIAL: NCT01085526
Title: Changes in Specific Immunoglobulin and Blood Basophil Activity During Subcutaneous Immunotherapy in Patients With Allergic Rhinitis Due to Grass Pollen Allergy - a Prospective Randomized Controlled Study
Brief Title: Changes in Specific Immunoglobulin and Blood Basophil Activity During Subcutaneous Immunotherapy in Allergic Rhinitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other); ALK-Abelló A/S (Industry); Lundbeck Foundation (Other)
Responsible Party: Principal Investigator, Pia Pedersen, MD, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BasoScit
Record Dates: First submitted 2010-03-10; First posted 2010-03-12 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2014-07

CONDITIONS: Allergic Rhinoconjunctivitis
Keywords: basophil activity; plasma cells; IgE; IgG1; IgG4; mast cells; IgE receptor; allergic rhinoconjunctivitis; grass pollen allergy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- alutard phl prat. treatment group (Active Comparator): 18 subjects receiving active treatment: basophil activity, plasma cells and immunoglobulins measured
  Interventions: Biological: Alutard phleum pratense subcutaneous immunotherapy; Drug: Alutard phl prat
- control group (No Intervention): control
- alutard phl.prat., treatment group2 (Active Comparator): basophil activity, basophil biology measured
  Interventions: Biological: Alutard phleum pratense subcutaneous immunotherapy; Drug: Alutard phl prat

INTERVENTIONS:
Biological: Alutard phleum pratense subcutaneous immunotherapy — standard regimen of SCIT
  Other Names: alutard phleum pratense; subcutaneous immunotherapy
  Arms: alutard phl prat. treatment group; alutard phl.prat., treatment group2
Drug: Alutard phl prat
  Other Names: Alutard 225, phleum pratense, ALK-abelló
  Arms: alutard phl prat. treatment group; alutard phl.prat., treatment group2

SUMMARY:
The trial is randomized prospective study to examine the effects of subcutaneous immunotherapy on the adaptive immune system. The trial includes 30 participants randomized to treatment or control group. The effect measures are changes in the basophil activity and biology as well as changes in plasma cells during and after treatment. Clinical outcome is assessed by QoL questionnaires and clinical testing.

Hypotheses:

* changes in plasma cells correlate to changes in immunoglobulins and effector cell responses
* the reduction of inflammation due to SCIT has influence on the effector cell responses
* changes in paraclinical measurements can be related to clinical findings

DETAILED DESCRIPTION:
The investigators are recruiting 30 participants, which are randomized to receive SCIT (24) or no treatment (6) The following will be measured

* the development of immunoglobulin response
* plasma cells under updosing phase
* changes in basophil activity under updosing and maintenance treatment
* subtyping of allergic sensitization
* clinical outcome and quality of life
* changes in mast cells in the nasal mucosa
* changes in the cell biology of the basophils

ELIGIBILITY:
Inclusion Criteria:

* rhinoconjunctivitis due to grass pollen allergy
* positive skin prick test and nasal allergen challenge test to grass pollen extract

Exclusion Criteria:

* severe comorbidity, severe asthma, pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-02; Primary Completion 2014-07 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
a significant decrease in basophil activity during and after treatment | every 3 weeks for 3 months, then 3 monthly for 3 years

SECONDARY OUTCOMES:
reduction in high affinity IgE receptor density on basophils and mast cells | at inclusion and at the end of study
  igE receptor density on basophils and mast cells from nasal mucosa
clinical outcome: reduction in the reaction to allergen challenge tests (skin and nose), significant better outcome in quality of life questionnaires and symptom/medication scores | once yearly for 4 years
  allergen challenging response
a significant increase in the number of plasma cells during up dosing | 5 times during the first 3 months of the study
a significant shift in specific immunoglobulins from IgE at start to IgG1 and IgG4 after treatment. allergen epitope specific IgE and IgG4 | every 3 months for 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Dahl, Prof, dr.med, Study Chair — Dept. of Respiratory Medicine, Århus University Hospital; Hans Juergen Hoffmann, assoc prof, Principal Investigator — Dept of Respiratory Medicine, Århus University Hospital; Johannes M Schmid, MD, Principal Investigator — Dept. of Respiratory Medicine, Aarhus University Hospital